CLINICAL TRIAL: NCT04683783
Title: RENACI Project: National Registry of Liver First Approach
Brief Title: National Registry of Liver First Approach
Acronym: RENACI
Status: Completed | Type: Observational
Sponsor: Hospital Miguel Servet (Other)
Collaborators: Spanish Association of Surgeons (AEC) (Other)
Responsible Party: Principal Investigator, Mario Serradilla, MD, FACS, MD, FACS, Hospital Miguel Servet
Other Study IDs: PI19/256
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Colonic Cancer; Rectal Cancer; Liver Metastases
Keywords: Liver first approach; Reverse strategy
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver metastases are present in 15-25% of patients with colorectal cancer at the time of diagnosis of the primary tumor, which is defined as synchronous liver metastases. Treatment for the potential cure of this disease includes surgical resection of both the primary tumor and liver metastases. The liver first approach was described by Mentha for patients with asymptomatic rectal tumors with with initially unresectable or borderline resectable liver metastases. There is little data in the scientific literature on how many patients scheduled for this strategy complete both surgeries and/or undergo the full chemo/radiation therapy.

DETAILED DESCRIPTION:
Liver metastases are present in 15-25% of patients with colorectal cancer at the time of diagnosis of the primary tumor, which is defined as synchronous liver metastases. Treatment for the potential cure of this disease includes surgical resection of both the primary tumor and liver metastases. However, due to the comorbidity or extent of the tumor disease, only a minority of patients are candidates for curative resections. When surgical treatment is indicated, different strategies can be used. In the classic strategy, the primary tumor is resected first, followed by surgery for metastases and, after that, adjuvant chemotherapy. More recently, simultaneous resection of primary and liver lesions has been used, mainly for limited liver disease without the need for large-volume liver resections. A third option is preoperative chemotherapy, followed by resection of liver metastases and surgery of the primary tumor in a second stage. This technique was initially described in 2006 by Mentha for patients with asymptomatic rectal tumors with initially unresectable or borderline resectable liver metastases. These patients were treated with neoadjuvant chemotherapy, followed by surgery for liver metastases, chemo/radiotherapy of the primary tumor, and second stage surgery. This is what is called surgery or reverse strategy (liver first approach in the Anglo-Saxon world). This strategy has the potential advantage of allowing resection of advanced liver disease in patients when the primary tumor is asymptomatic. Advanced liver disease is the leading cause of mortality in these patients. Subsequently, this strategy has been used in colorectal tumors of any location with synchronous metastases. No clear advantage or disadvantage has been demonstrated with any of the three strategies in terms of long-term survival. There is also no prospective randomized clinical trial comparing classical with reverse strategy.

Most of the previous studies that evaluated this strategy only included patients with liver resection, not the primary one. Therefore, there is little data in the scientific literature on how many patients scheduled for this strategy complete both surgeries and/or undergo the full chemo/radiation therapy. The potential advantage of this strategy is the possibility of rescuing more patients with colorectal cancer liver metastases, thus increasing survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 year old.
* Scheduled surgery for colorectal cancer with synchronous liver metastases using the liver first approach.
* ASA score I-III.
* They have signed the informed consent.

Exclusion Criteria:

* Patients under 18 year old.
* ASA ≥ IV.
* Urgent surgery.
* Patients who have not signed the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients operated on in the participating Spanish centers with colorectal cancer and synchronous liver metastases who underwent a liver first approach during the study period and that meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who complete the entire cycle | 90 days
  Percentage of patients who complete the cycle: neoadjuvant chemotherapy - liver surgery - CT / RT of the primary - surgery of the primary tumor

SECONDARY OUTCOMES:
Mortality rate | 90 days
  Postoperative mortality including liver surgery and primary tumor
Morbidity rate | 90 days
  Postoperative morbidity including liver surgery and primary tumor (all type of postoperative complications)

CONTACTS AND LOCATIONS:
Locations (1):
- Mario Serradilla Martín, Zaragoza, Spain

REFERENCES:
- [Result] Jegatheeswaran S, Mason JM, Hancock HC, Siriwardena AK. The liver-first approach to the management of colorectal cancer with synchronous hepatic metastases: a systematic review. JAMA Surg. 2013 Apr;148(4):385-91. doi: 10.1001/jamasurg.2013.1216. PMID 23715907
- [Result] de Jong MC, van Dam RM, Maas M, Bemelmans MH, Olde Damink SW, Beets GL, Dejong CH. The liver-first approach for synchronous colorectal liver metastasis: a 5-year single-centre experience. HPB (Oxford). 2011 Oct;13(10):745-52. doi: 10.1111/j.1477-2574.2011.00372.x. Epub 2011 Sep 5. PMID 21929676
- [Result] Lam VW, Laurence JM, Pang T, Johnston E, Hollands MJ, Pleass HC, Richardson AJ. A systematic review of a liver-first approach in patients with colorectal cancer and synchronous colorectal liver metastases. HPB (Oxford). 2014 Feb;16(2):101-8. doi: 10.1111/hpb.12083. Epub 2013 Mar 19. PMID 23509899
- [Result] Tsoulfas G, Pramateftakis MG. Management of rectal cancer and liver metastatic disease: which comes first? Int J Surg Oncol. 2012;2012:196908. doi: 10.1155/2012/196908. Epub 2012 Jun 20. PMID 22778934
- [Result] Mentha G, Majno PE, Andres A, Rubbia-Brandt L, Morel P, Roth AD. Neoadjuvant chemotherapy and resection of advanced synchronous liver metastases before treatment of the colorectal primary. Br J Surg. 2006 Jul;93(7):872-8. doi: 10.1002/bjs.5346. PMID 16671066
- [Result] Mayo SC, Pulitano C, Marques H, Lamelas J, Wolfgang CL, de Saussure W, Choti MA, Gindrat I, Aldrighetti L, Barrosso E, Mentha G, Pawlik TM. Surgical management of patients with synchronous colorectal liver metastasis: a multicenter international analysis. J Am Coll Surg. 2013 Apr;216(4):707-16; discussion 716-8. doi: 10.1016/j.jamcollsurg.2012.12.029. Epub 2013 Feb 21. PMID 23433970
- [Result] Adam R, De Gramont A, Figueras J, Guthrie A, Kokudo N, Kunstlinger F, Loyer E, Poston G, Rougier P, Rubbia-Brandt L, Sobrero A, Tabernero J, Teh C, Van Cutsem E; Jean-Nicolas Vauthey of the EGOSLIM (Expert Group on OncoSurgery management of LIver Metastases) group. The oncosurgery approach to managing liver metastases from colorectal cancer: a multidisciplinary international consensus. Oncologist. 2012;17(10):1225-39. doi: 10.1634/theoncologist.2012-0121. Epub 2012 Sep 7. PMID 22962059
- [Result] Adam R, de Gramont A, Figueras J, Kokudo N, Kunstlinger F, Loyer E, Poston G, Rougier P, Rubbia-Brandt L, Sobrero A, Teh C, Tejpar S, Van Cutsem E, Vauthey JN, Pahlman L; of the EGOSLIM (Expert Group on OncoSurgery management of LIver Metastases) group. Managing synchronous liver metastases from colorectal cancer: a multidisciplinary international consensus. Cancer Treat Rev. 2015 Nov;41(9):729-41. doi: 10.1016/j.ctrv.2015.06.006. Epub 2015 Jun 30. PMID 26417845
- [Result] Ihnat P, Vavra P, Zonca P. Treatment strategies for colorectal carcinoma with synchronous liver metastases: Which way to go? World J Gastroenterol. 2015 Jun 14;21(22):7014-21. doi: 10.3748/wjg.v21.i22.7014. PMID 26078580
- [Result] Waisberg J, Ivankovics IG. Liver-first approach of colorectal cancer with synchronous hepatic metastases: A reverse strategy. World J Hepatol. 2015 Jun 18;7(11):1444-9. doi: 10.4254/wjh.v7.i11.1444. PMID 26085905
- [Result] Sturesson C, Valdimarsson VT, Blomstrand E, Eriksson S, Nilsson JH, Syk I, Lindell G. Liver-first strategy for synchronous colorectal liver metastases - an intention-to-treat analysis. HPB (Oxford). 2017 Jan;19(1):52-58. doi: 10.1016/j.hpb.2016.10.005. Epub 2016 Nov 9. PMID 27838252
- [Result] Regimbeau JM, Cosse C, Kaiser G, Hubert C, Laurent C, Lapointe R, Isoniemi H, Adam R. Feasibility, safety and efficacy of two-stage hepatectomy for bilobar liver metastases of colorectal cancer: a LiverMetSurvey analysis. HPB (Oxford). 2017 May;19(5):396-405. doi: 10.1016/j.hpb.2017.01.008. Epub 2017 Mar 23. PMID 28343889